CLINICAL TRIAL: NCT07163832
Title: Retrospective Single-center Study of the Cohort of Transgender Patients Who Began Medical Support Before the Age of 18 at the Strasbourg University Hospital
Brief Title: Retrospective Study of the Cohort of Transgender Patients Who Began Medical Support Before the Age of 18
Acronym: TRANS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9688
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Endocrinology
Keywords: Pediatric endocrinology; Child Psychiatry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gender incongruence is characterized by a marked and persistent incongruity between the gender with which a person identifies and their assigned sex. Behaviors and preferences that vary by sex do not, in and of themselves, justify the assignment of diagnoses in this group.

ELIGIBILITY:
Inclusion Criteria:

* Minor patient (≥18 years old)
* First-time patient for transgender issues at the Strasbourg University Hospital in child psychiatry and/or pediatric endocrinology (in at least one of the two departments)
* Patient (and/or their legal representative) who has not expressed opposition to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Patient (and/or their representative) who has expressed opposition to the reuse of their data for scientific research purposes.
* Patient aged over 18 at the first consultation
* Patient with insufficient data

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor patient (≥18 years old) who has been consulted for the first time for transgender issues at the Strasbourg University Hospital in child psychiatry and/or pediatric endocrinology (in at least one of the two departments)
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Retrospective descriptive study of the population of transgender minors receiving medical support at the Strasbourg University Hospital | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Service de pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France